CLINICAL TRIAL: NCT01394380
Title: Effects of a Reduction of Sweetened Beverages Consumption in Overweight High Consumers on Cardiometabolic Risk Factors
Brief Title: Reduction of Sweetened Beverages and Intrahepatic Fat
Acronym: REDUCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, professor of physiology, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 171/11
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Obesity; Dyslipidemia; Metabolic Syndrome
Keywords: sugar; sweetened beverages; hepatic steatosis; visceral obesity; metabolic syndrome
MeSH Terms: conditions — Obesity; Dyslipidemias; Metabolic Syndrome; Fatty Liver; Obesity, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- artificially sweetened beverages (Experimental): subjects will be required to consume only artificially-sweetened sodas, water, tea or coffee
  Interventions: Other: artificially sweetened sodas
- regular sodas (No Intervention): subjects will continue their usual consumption of sweetened sodas

INTERVENTIONS:
Other: artificially sweetened sodas — subjects will be allowed unlimited consumption of calorie-free, artificially-sweetened sodas, water, tea or coffee
  Arms: artificially sweetened beverages

SUMMARY:
The study will enroll 68 overweight male and female subjects with a high (> 2 3dl-can soda/day) consumption of sweetened beverage per day. After a run-in period of 4 weeks, subjects will be randomized to either a 12-week intervention arm in which sweetened beverages will be replaced by artificially sweetened, calorie-free beverages, or to a control arm. The following measurements will be performed at the end of the run-in period and at the end of the intervention period

* intrahepatic fat concentration
* visceral fat volume
* changes in day-long metabolic profile from baseline(plasma glucose, insulin, and triglyceride concentrations)
* changes in food intake and daily energy, carbohydrate and sugars intake from baseline

ELIGIBILITY:
Inclusion Criteria:

* gender male or female
* body mass index (BMI) > 27 kg/m2 consumption of > 2 3dl-can regular soda/day
* low to moderate physical activity (< 60 min walking/day; < 3 exercise session/week

Exclusion Criteria:

* diabetes mellitus
* liver, kidney or heart disease
* any current drug treatment
* contra-indications to MR examination (pacemaker, foreign bodies,etc)
* pregnancy or planned pregnancy
* active weight gain or weight loss (weight change > 4 kg in the past 12 months)
* consumption of drugs or illicit substances
* consumption of more than 10g alcohol/day
* vegetarians or subjects on special diets

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
changes in intrahepatic fat concentration | at the end of run-in and after 12 weeks intervention/control
  intrahepatic fat content measured by 1H-MRS

SECONDARY OUTCOMES:
changes in visceral fat volume | at the end of run-in and after 12 weeks of intervention/control
  Visceral fat volume measured by MRI
changes in day-long metabolic profile | at the end of run-in and after 12 weeks of intervention/control
  Plasma glucose, insulin, non-esterified fatty acids, and triglycerides will be measured at 2-hourly intervals between 7:00 am and 5:00 pm. Participants will be fed standardized meals and either sweetened or artificially-sweetened beverages according to randomization
changes in food intake from baseline | at the end of the run-in period and after 6, and 12 weeks of intervention/control
  Total energy intake, total carbohydrate intake, and total sugars intake will be evaluated by 3-day food record

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, MD, Principal Investigator — Department of Physiology, University of Lausanne
Locations (1):
- Clinical Research Center, CHUV, Lausanne, Canton of Vaud, Switzerland